CLINICAL TRIAL: NCT02229097
Title: Clinical Efficacy of Coordinated Boluses in Type 1 Diabetic Patients Treated With Insulin Pumps: a Multicentric, Randomised, Cross Over Study
Brief Title: Efficacy of Coordinated Insulin Boluses in Type 1 Diabetic Patients
Acronym: COBOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13 7029 08; 2014-000969-47 (EudraCT Number); 13-074 (Other Grant/Funding Number: French Ministry of Health, PHRC 2013)
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal then Coordinated (Experimental): normal bolus during 2 weeks then coordinated bolus during 2 weeks
  Interventions: Drug: Normal bolus; Drug: Coordinated bolus
- Coordinated then Normal (Experimental): coordinated bolus during 2 weeks then normal bolus during 2 weeks
  Interventions: Drug: Normal bolus; Drug: Coordinated bolus

INTERVENTIONS:
Drug: Normal bolus — During the "normal bolus" period, the bolus will be adjusted to the carbohydrate content of each meal and injected immediately. The basal rate will remain at a normal level during the 3 hours postprandial period
Drug: Coordinated bolus — The basal rate will be reduced at a rate of 0.1 U/h during the 3 h postprandial period. The insulin subtracted of the basal rate will be added to the normal bolus calculated for the meal and injected immediately.

SUMMARY:
A recent study suggests that, in Type 1 Diabetes (T1D) patients treated by insulin pumps, a better coordination of meal boluses and post prandial basal rate could reduce the importance of postprandial hyperglycaemias without increasing the risk of delayed hypoglycaemias.

The aim of the investigators study is to assess if these results are confirmed in a clinical trial.

The aim of this study is to compare the efficacy of coordinated boluses versus normal boluses on postprandial glycaemic control of T1D patients treated with continuous subcutaneous insulin infusion.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* with confirmed Negative C-peptide or diabetes duration>5 years
* Treated by external insulin pump and rapid insulin analog for more than 3 months
* using a Medtronic Paradigm Real-Time or Veo™ model
* Educated to and practicing functional insulin treatment and carbohydrate counting for more than 3 months
* Able to use the "basal temp" and "glycaemia reminder" functions of their pump
* Basal infusion rate ≥ 0,5 Unit/h
* Self-monitoring of blood glucose frequency > 4/days
* Aware of hypoglycaemia

Exclusion Criteria:

* known impaired renal function (creatinin clearance <60ml/min)
* Gastroparesis
* Serious or instable disease likely to induce a glycaemic control deterioration - treatment with corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
postprandial glycaemia | 2 hours after eating during 4 weeks
  measured by Self Monitoring of Blood Glucose

SECONDARY OUTCOMES:
adverse events | Throughout the study (4 weeks)
severe hypoglycaemia frequency | Throughout the study (4 weeks)
insulin doses | basal rate and boluses
mean glycaemia | before eating and 2 hours after eating during 4 weeks
  data from Self Monitoring of Blood Glucose
standard deviation of glycaemia | before eating and 2 hours after eating during 4 weeks
  data from Self Monitoring of Blood Glucose
frequency of glycaemia < or = 60mg/dl | before eating and 2 hours after eating during 4 weeks
  data from Self Monitoring of Blood Glucose
frequency of glycaemia between 61-140mg/dl | before eating and 2 hours after eating during 4 weeks
  data from Self Monitoring of Blood Glucose
frequency of glycaemia >140mg/dl | before eating and 2 hours after eating during 4 weeks
  data from Self Monitoring of Blood Glucose
mean glycemia | Throughout the day during 4 weeks
  data from Continue Glycemia Monitoring
standard deviation | Throughout the day during 4 weeks
  data from Continue Glycemia Monitoring
time spent within glucose range < or = 60mg/dl | Throughout the day during 4 weeks
  data from Continue Glycemia Monitoring
time spent within glucose range between 61-140mg/dl | Throughout the day during 4 weeks
  data from Continue Glycemia Monitoring
time spent within glucose range mg/dl | Throughout the day during 4 weeks
  data from Continue Glycemia Monitoring
fructosamine | day 1
fructosamine | day 1 + 2 weeks
fructosamine | day 1 + 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Melki, Doctor, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - University Hospital Toulouse Rangueil, Toulouse, Haute Garonne
  - Saint-André Hospital, Bordeaux
  - Lapeyronie Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bondia J, Dassau E, Zisser H, Calm R, Vehi J, Jovanovic L, Doyle FJ 3rd. Coordinated basal-bolus infusion for tighter postprandial glucose control in insulin pump therapy. J Diabetes Sci Technol. 2009 Jan;3(1):89-97. doi: 10.1177/193229680900300110. PMID 20046653
- [Background] A. Farret, B. Catargi, J.P. Riveline, V. Melki, P. Schaepelynck, A. Sola, B. Guerci, H. Bertet, T. Mura, H. Chevassus, E. Renard : Étude randomisée contrôlée en cross-over comparant les effets sur le contrôle glycémique des bolus immédiats et combinés chez des patients diabétiques de type 1 traités par pompe à insuline portable. Diabetes & Metabolism, Volume 38, Supplement 2, March 2012, Page A6
- [Background] Druet C, Roudier C, Romon I, Assogba F, Bourdel-Marchasson I, et al. Échantillon national témoin représentatif des personnes diabétiques, Entred 2007-2010.
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Etude Jubilé. SFD 2013
- [Background] Pickup J, Mattock M, Kerry S. Glycaemic control with continuous subcutaneous insulin infusion compared with intensive insulin injections in patients with type 1 diabetes: meta-analysis of randomised controlled trials. BMJ. 2002 Mar 23;324(7339):705. doi: 10.1136/bmj.324.7339.705. PMID 11909787
- [Background] Mudaliar SR, Lindberg FA, Joyce M, Beerdsen P, Strange P, Lin A, Henry RR. Insulin aspart (B28 asp-insulin): a fast-acting analog of human insulin: absorption kinetics and action profile compared with regular human insulin in healthy nondiabetic subjects. Diabetes Care. 1999 Sep;22(9):1501-6. doi: 10.2337/diacare.22.9.1501. PMID 10480516
- [Background] Directive pour la gestion de la glycémie post prandiale, IDF 2007 http://www.idf.org/webdata/docs/French_GMPG Final 110108.pdf
- [Background] Melki.v, Cazals.l : Impact de la coordination des bolus et du débit de base sur le contrôle des glycémies postprandiales chez des diabétiques de type 1 traités par pompe externe (étude pilote). Poster accepté SFD 2014